CLINICAL TRIAL: NCT06433648
Title: Understanding How Powered Componentry Impacts K2-Level Transfemoral Amputee Gait
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Levi Hargrove, Scientific Chair, Center for Bionic Medicine, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STU00217960
Record Dates: First submitted 2024-05-16; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Amputation; Amputation, Traumatic; Amputation of Knee; Amputation; Traumatic, Limb
MeSH Terms: conditions — Amputation, Traumatic

STUDY DESIGN:
Intervention Model Description: The goal of this study is to understand how providing power at the knee or ankle individually, or providing power at both the knee and ankle, impacts ambulation for transfemoral amputees with limited community mobility.
  Aim 1: measure functional performance of transfemoral ambulators when using a commercially available passive microprocessor knee prosthesis (Ottobock Cleg/Ottobock foot) or a powered knee and ankle prosthesis (SRALab Hybrid Knee and SRAlab Polycentric Powered Ankle.
  Aim 2: Participants will be evaluated on the contribution of adding power at the knee only or the ankle only.
  Aim 3: The investigators will evaluate the functional performance after intensive clinical gait training on the powered knee and ankle prosthesis (SRALab Hybrid Knee and SRALab Polycentric Powered Ankle).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Transfemoral Amputee participants: Ottobock Cleg4 + Ottobock foot; Hybrid Knee + Polycentric Ankle (Active Comparator): Participant is fit with the commercially available device (Ottobock Cleg 4/Ottobock foot), they will receive standard of care clinical training for 3-4 sessions over 4 weeks, plus 1 session for outcome assessments.
  Participant is then fit with the SRALAB Hybrid knee and SRALAB Polycentric Ankle prosthesis, they again will receive clinical training for 3-4 sessions over 4 weeks, plus 1 session for outcome assessments.
  Interventions: Device: Ottobock CLeg4 + Ottobock foot; Device: SRALAB Hybrid Knee + Polycentric Ankle
- Transfemoral Amputee participants: Ottobock CLeg4 + Polycentric Ankle, Hybrid Knee + Passive Ankle (Experimental): For this arm, transfemoral amputees will participate in an AB/BA randomized crossover study.
  Before each arm of the cross-over, baseline data will be taken with the Ottobock Cleg 4/Ottobock foot or their clinically prescribed microprocessor knee unit/foot.
  Condition A is CLeg + Polycentric Ankle
  Condition B is SRALab Hybrid knee + Passive Ankle
  Subjects will participate in 2 sessions over 2 weeks, each lasting 2-3 hours to have the device tuned for the specific condition (A or B). On the third week, they will participate in 2 visits to complete functional outcome measures, biomechanical and metabolic assessments. They will then switch conditions, and repeat the protocol for the second condition.
  There will not be a washout period between conditions, but subjects will complete outcome measures with the Ottobock Cleg 4/Ottobock foot or their clinically prescribed microprocessor knee unit/foot prior to each arm of the crossover to obtain baseline data.
  Interventions: Device: SRALAB Hybrid Knee + Passive Ankle; Device: Ottobock CLeg 4 + Polycentric Ankle
- Transfemoral Amputee participants: SRALAB Hybrid knee + Polycentric Ankle, Ottobock Cleg4 + OB foot (Experimental): During this arm, participants will receive intensive clinical training with the SRALAB Hybrid knee + Polycentric Ankle twice per week over 8 weeks, lasting 2-3 hours. Training will include patient-driven therapy to achieve participants' individual therapy goals, functional mobility and community skills.
  At the end of the 8-week training period, subjects will complete the same set of functional outcome measures, biomechanical and metabolic assessments in previous arms.
  To complete this arm, participants will again complete training and outcome measures with the Ottobock Cleg4/Ottobock or their clinically prescribed microprocessor knee unit/foot over 3 visits.
  Interventions: Device: Ottobock CLeg4 + Ottobock foot; Device: SRALAB Hybrid Knee + Polycentric Ankle

INTERVENTIONS:
Device: Ottobock CLeg4 + Ottobock foot — Commercially available Ottobock CLeg 4 microprocessor knee unit and Ottobock foot.
  Arms: Transfemoral Amputee participants: Ottobock Cleg4 + Ottobock foot; Hybrid Knee + Polycentric Ankle; Transfemoral Amputee participants: SRALAB Hybrid knee + Polycentric Ankle, Ottobock Cleg4 + OB foot
Device: SRALAB Hybrid Knee + Polycentric Ankle — Experimental powered prosthesis: SRALAB Hybrid Knee and powered polycentric ankle.
  Arms: Transfemoral Amputee participants: Ottobock Cleg4 + Ottobock foot; Hybrid Knee + Polycentric Ankle; Transfemoral Amputee participants: SRALAB Hybrid knee + Polycentric Ankle, Ottobock Cleg4 + OB foot
Device: SRALAB Hybrid Knee + Passive Ankle — Experimental powered prosthesis: SRALAB Hybrid Knee and passive ankle.
  Arms: Transfemoral Amputee participants: Ottobock CLeg4 + Polycentric Ankle, Hybrid Knee + Passive Ankle
Device: Ottobock CLeg 4 + Polycentric Ankle — Commercially available Ottobock CLeg 4 prosthetic knee and SRALAB powered polycentric ankle.
  Arms: Transfemoral Amputee participants: Ottobock CLeg4 + Polycentric Ankle, Hybrid Knee + Passive Ankle

SUMMARY:
The goal of this study is to understand how providing power at the knee or ankle individually, or providing power at both the knee and ankle, impacts ambulation for K2 level transfemoral amputees.

Aim 1: measure functional performance of K2 level ambulators when using a commercially available passive microprocessor knee prosthesis (Ottobock Cleg/Ottobock foot) or a powered knee and ankle prosthesis (SRALab Hybrid Knee and SRAlab Polycentric Powered Ankle.

Aim 2: Participants will be evaluated on the contribution of adding power at the knee only or the ankle only.

Aim 3: The investigators will evaluate the functional performance after intensive clinical gait training on the powered knee and ankle prosthesis (SRALab Hybrid Knee and SRALab Polycentric Powered Ankle).

Our hypothesis is that providing powered componentry will improve function and that intensive training will magnify those improvements.

DETAILED DESCRIPTION:
Amputation of the lower limb causes profound disability, significantly limiting mobility, independence, and the ability to pursue employment or leisure activities. Nearly 90% of all lower limb amputations in the United States occur in older persons, mostly due to vascular disease, and this population is expected to triple by 2050. After lower limb loss, individuals walk more slowly and more asymmetrically are less stable, and expend more metabolic energy during walking than persons with intact limbs. Even when using state-of-the-art microprocessor-controlled prostheses (typically a microprocessor knee with a passive ankle), persons with transfemoral amputations expend approximately 60% more energy than able-bodied individuals during ambulation. In addition to the physical limitations caused by the amputation, the increased energy requirements affect performance of everyday activities, including getting up out of a chair or off the toilet, or stepping up or down a curb.

Most commercially available prosthetic legs are passive. The movement of a passive prosthetic joint relies on the properties of its mechanical components, such as hydraulic or pneumatic valves or sliding joints, together with compensatory adjustments made by the user. Since these computerized prostheses are passive, the user cannot efficiently negotiate stairs, an incline, or the numerous other functions that require net knee and/or ankle power.

Powered prostheses can actively generate joint torque, allowing easy and efficient performance of more demanding activities, such as ascending stairs and hills. Powered knees and ankles, may allow for better outcomes in both older and younger individuals with transfemoral amputation; this powered componentry may enable more energy efficient walking, allow users to stand up from a seated position with ease, and enable them to walk across more challenging terrains-such as up and down hills, ramps, and stairs-safely and with more normal and symmetric gait kinematics and kinetics.

This study will demonstrate the functional benefits of adding power at an individual joint. This knowledge will be critical for prioritizing future device development and will provide valuable information for clinicians and individuals on selecting appropriate componentry for transfemoral K2 amputees.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-95
* A unilateral transfemoral amputation
* At least 6 months since definitive prosthesis fitting
* Able to walk 50 meters (55 yards) with a prosthesis without the assistance of another person.
* Medically cleared by physician to participate in study
* English speaking

Exclusion Criteria:

* Weight greater than 250 pounds
* Significant new injury that would prevent use of a prosthesis: The ability to consistently wear a prosthesis and perform activities of daily living and specific performance tasks is necessary to evaluate the relative benefits of the interventions.
* Cognitive impairment sufficient to adversely affect understanding of or compliance with study requirements, ability to communicate experiences, or ability to give informed consent: The ability to understand and comply with requirements of the study is essential in order for the study to generate useable, reliable data. The ability to obtain relevant user feedback through questionnaires and informal discussion adds significant value to this study.
* Significant other comorbidity: Any other medical issues or injuries that would preclude completion of the study, use of the prostheses, or that would otherwise prevent acquisition of useable data by researchers.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Amputee Mobility Predictor with Prosthesis (AMPRO) score | Completed at visit during week 5, week 10, week 11, week 14, week 15, week 18, week 35 and week 38.
  The AMPRO measures the ambulatory potential of lower limb amputees. It is used to assess functional mobility through a standardized sequence of mobility tests while using a prosthesis. Individual tasks are scored and combined, resulting in a total assessment score out of a possible 47; the minimum score is zero. Higher scores indicate better mobility.
  The AMPPRO is a reliable performance measure that has been validated for those with lower limb loss; it measures several functional mobility tasks that are needed during activities of daily living; it has been used to identify limitations in prosthetic mobility, including tasks that require both vertical mobility (sit/stand), horizontal mobility (walking), and balance. The AMPPRO scores have been shown to differentiate between Medicare K-levels and to provide information to guide therapeutic exercise techniques and document change after clinical instruction.

SECONDARY OUTCOMES:
6 Minute Walk Test (6MWT) | Completed at visit during week 5, week 10, week 11, week 14, week 15, week 18, week 35 and week 38.
  The 6 minute walk test (6MWT) assesses distance walked over 6 minutes as a sub-maximal test of aerobic capacity/endurance.
Timed Up and Go (TUG) | Completed at visit during week 5, week 10, week 11, week 14, week 15, week 18, week 35 and week 38.
  The Timed Up and Go Test (TUG) assesses mobility, balance, walking ability, and fall risk in older adults.
Four Square Step Test (FSST) | Completed at visit during week 5, week 10, week 11, week 14, week 15, week 18, week 35 and week 38.
  A test of dynamic balance and coordination that clinically assesses the participant's ability to step over objects forward, sideways, and backwards.
Metabolic Testing | Completed at visit during week 5, week 10, week 11, week 14, week 15, week 18, week 35 and week 38
  Subjects will be instrumented with the COSMED® K5 system (COSMED, Rome, Italy). Baseline metabolic data prior to each walking bout will be recorded for 2 minutes of sitting and quiet rest. Metabolic data will then be collected during 6 minutes of walking at a constant self-selected walking velocity on a treadmill. After each walking bout, subjects will rest for 20 minutes to allow their heart rate to return to their baseline level.

CONTACTS AND LOCATIONS:
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

REFERENCES:
- [Background] Ziegler-Graham K, MacKenzie EJ, Ephraim PL, Travison TG, Brookmeyer R. Estimating the prevalence of limb loss in the United States: 2005 to 2050. Arch Phys Med Rehabil. 2008 Mar;89(3):422-9. doi: 10.1016/j.apmr.2007.11.005. PMID 18295618
- [Background] Gailey RS, Wenger MA, Raya M, Kirk N, Erbs K, Spyropoulos P, Nash MS. Energy expenditure of trans-tibial amputees during ambulation at self-selected pace. Prosthet Orthot Int. 1994 Aug;18(2):84-91. doi: 10.3109/03093649409164389. PMID 7991365
- [Background] Hafner BJ, Sanders JE, Czerniecki J, Fergason J. Energy storage and return prostheses: does patient perception correlate with biomechanical analysis? Clin Biomech (Bristol). 2002 Jun;17(5):325-44. doi: 10.1016/s0268-0033(02)00020-7. PMID 12084537
- [Background] Burger H, Marincek C. The life style of young persons after lower limb amputation caused by injury. Prosthet Orthot Int. 1997 Apr;21(1):35-9. doi: 10.3109/03093649709164528. PMID 9141124
- [Background] Fey NP, Simon AM, Young AJ, Hargrove LJ. Controlling Knee Swing Initiation and Ankle Plantarflexion With an Active Prosthesis on Level and Inclined Surfaces at Variable Walking Speeds. IEEE J Transl Eng Health Med. 2014 Jul 25;2:2100412. doi: 10.1109/JTEHM.2014.2343228. eCollection 2014. PMID 27170878
- [Background] Adamczyk PG, Kuo AD. Mechanisms of Gait Asymmetry Due to Push-Off Deficiency in Unilateral Amputees. IEEE Trans Neural Syst Rehabil Eng. 2015 Sep;23(5):776-85. doi: 10.1109/TNSRE.2014.2356722. Epub 2014 Sep 12. PMID 25222950